CLINICAL TRIAL: NCT03245905
Title: Study of Chidamide as a Single-agent Treatment for Patients With Relapse or Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Study of Chidamide as a Single-agent Treatment for Patients With Relapse or Refractory B-NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Chief, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-B09
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental): Chidamide should be given at a fixed time with fixed dosage
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide 30mg orally BIW. Treatment cycles are repeated every 3 weeks.The maximum duration of treatment is 2 years.
  Other Names: epidaza

SUMMARY:
This is a prospective phase II clinical trial to observe the efficacy and safety of Chidamide as a single-agent treatment in patients with relapsed or refractory B-cell Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
Patients with relapsed /refractory aggressive B cell lymphoma usually have a poor prognosis. These patients cannot be treated successfully or tolered with the conventional chemotherapy. Epigenetic changes in B-cell lymphoma. Thus, epigenetic agents may offer potential improvment of clinical outcomes. Chidamide is a new type of oral histone deacetylase inhibitor. Our exploratory research found that Chidamide was effect in some relapsed /refractory B cell lymphoma patients

. Thus, we will evaluate the efficacy and safety of Chidamide in the patients with aggressive relapsed refractory B cell lymphoma failed from second line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as B-cell Non-Hodgkin's Lymphoma (NHL) according to "2008 WHO classification of tumors of haematopoietic and lymphoid tissues", including Diffuse Large B-Cell Lymphoma (DLBCL), Mantle Cell Lymphoma (MCL), transformed indolent lymphoma (TL), and other subtypes that investigators consider to be appropriate to be enrolled;
2. Patients achieved CR or PR in previous cytotoxic chemotherapy, and relapsed later than 6 months after remission;
3. Patients with DLBCL, FL grade3, MALT, LPL and SLL received at least two chemotherapy regimens, and Patients with FL grade1-2 received at least three chemotherapy regimens;
4. At least one measurable lesion with a longest diameter >1.5cm or a short axis >1.0cm;
5. Age18-75 years;
6. ECOG performance status 0-2;
7. Life expectancy no less than 3 months;
8. Functions within 7 days prior to enrollment: Blood routine test: Hb ≥ 80g/L, absolute neutrophil count ≥1.5 × 109/L, platelet ≥60 × 109/L; Total bilirubin ≤ 1.5 times of normal maximum, ALT/AST≤ 2.5 times of normal maximum, for patients with liver metastasis ALT/AST≤ 5 times of normal maximum; serum creatinin≤1.5 times of normal maximum or CCr≥ 60ml/min;
9. LVEF ≥ 50% by echocardiography;
10. Contraception during and 4 weeks after the study for patients at child bearing age;
11. Patients have signed the Informed Consent Form.

Exclusion Criteria:

1. Patients received Chidamide treatment within 6 months prior to enrollment;
2. Patients with Burkitt Lymphoma, B-lymphoblastic lymphoma, central nervous system lymphoma and HIV-Associated Lymphoma;
3. Patients with a "currently active" second malignancy;
4. Patients not recovered from non-hematologic toxicities within 4 weeks prior to enrollment due to chemotherapy, radiation and immunotherapy;
5. Patients receiving or received corticosteroids within 2 weeks prior to enrollment;
6. Patients with cumulative life time dose of Doxorubicin > 450mg/m2;
7. Patients who have been treated with any investigational drug within 4 weeks prior to enrollment;
8. Women during pregnancy or lactation;
9. Patients with active infection, medical conditions, or mental disorders;
10. Patients with active infection of HBV, HCV or HIV;
11. Congestive heart failure (NYHA grade III/IV), myocardial infarction within 6 months, QTc elongation with clinical significance (≥480ms), hypertension BP≥150/100 mmHg and symptomatic coronary heart disease that require treatment;
12. Patients with drug abuse, long term alcoholism that may impact the results of the trial;
13. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | every 6 weeks until 2 years after last patient's enrollment
  Overall response was determined on the basis of investigator assessments according to lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET.

SECONDARY OUTCOMES:
progression-free survival（PFS） | every 6 weeks until 2 years after last patient's enrollment
  The time between the start of randomization and the progression of the tumor (any aspect) or (for any reason) death
overall survival（OS） | every 6 weeks until 2 years after last patient's enrollment
  Time from randomization to death for any reason Time from randomization to death for any reason Time from randomization to death for any reason Time from randomization to death for any reason
Percentage of Participants With Adverse Events (AEs) | Up to 36 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No